CLINICAL TRIAL: NCT01483742
Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics and Antiviral Activity of Ritonavir-Boosted DANOPREVIR and RO5024048 in Different Combinations in Null Responder or Treatment Naïve Patients With Chronic Hepatitis C and Compensated Cirrhosis
Brief Title: A Study of Ritonavir-Boosted Danoprevir and RO5024048 in Different Combinations in Null Responder or Treatment-Naïve Patients With Chronic Hepatitis C and Compensated Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP27946; 2011-004129-28 (EudraCT Number)
Record Dates: First submitted 2011-11-30; First posted 2011-12-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — danoprevir; peginterferon alfa-2a; Ribavirin; Ritonavir

ARMS (2):
- Combination without RO5024048 (Experimental): Ritonavir-boosted danoprevir in combination with Pegasys (peginterferon alfa-2a) and ribavirin in treatment-naïve patients
  Interventions: Drug: danoprevir; Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin; Drug: ritonavir
- Combination with RO5024048 (Experimental): RO5024048 added to the combination treatment (ritonavir-boosted danoprevir in combination with Pegasys [peginterferon alfa-2a] and ribavirin) in prior null responder patients
  Interventions: Drug: RO5024048; Drug: danoprevir; Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin; Drug: ritonavir

INTERVENTIONS:
Drug: RO5024048 — 1000 mg orally bid, 24 weeks
  Arms: Combination with RO5024048
Drug: danoprevir — 100 mg orally bid, 24 weeks
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg weekly, 24 weeks
Drug: ribavirin — 1000-1200 mg/kg/day orally in two divided doses, 24 weeks
Drug: ritonavir — 100 mg orally bid, 24 weeks

SUMMARY:
This open-label, parallel cohort study will evaluate the safety, pharmacokinetics and antiviral activity of ritonavir-boosted danoprevir in combination with Pegasys (peginterferon alfa-2a) and ribavirin in treatment-naïve patients, and with RO5024048 added to the combination treatment in prior null responder patients with chronic hepatitis C genotype 1 or 4 and compensated cirrhosis. All patients will receive danoprevir 100 mg orally twice daily (bid) , ritonavir 100 mg orally bid, Pegasys 180 mcg subcutaneously weekly and ribavirin 1000-1200 mg/kg/day orally. Prior non-responders will receive RO5024048 1000 mg orally bid additionally. Anticipated time on study treatment is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 to 65 years of age inclusive
* Chronic hepatitis C, genotype 1 or 4
* Cohort 1: Treatment-naïve for hepatitis C
* Cohort 2: Prior null responder to treatment with approved doses of pegylated interferon plus ribavirin
* Liver biopsy confirming cirrhosis
* Compensated cirrhosis (Child-Pugh A)

Exclusion Criteria:

* Pregnant or lactating women or male partners of women who are pregnant
* History or presence of decompensated liver disease (ascites, hepatic encephalopathy, hepatocellular carcinoma, or bleeding esophageal varices)
* Cohort 2: Patients who discontinued previous pegylated interferon plus ribavirin treatment due to reasons other than null response
* History of clinically significant cardiovascular or cerebrovascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 48 weeks
Pharmacokinetics (PK): Area under the concentration-time curve (AUC) | Intensive PK sample collection during initial 2 week dosing period, followed by routine sampling during treatment up to Week 24
Antiviral activity: Hepatitis C virus (HCV) RNA levels assessed by Roche COBAS Taqman HCV Test | 48 weeks

SECONDARY OUTCOMES:
Emergence of viral resistance: HCV RNA gene sequence variations | From baseline to Week 48
Virologic response: HCV RNA levels | approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- United States (14):
  - Birmingham, Alabama
  - Anaheim, California
  - Coronado, California
  - La Jolla, California
  - Long Beach, California
  - DeLand, Florida
  - Miami, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - New Orleans, Louisiana
  - Detroit, Michigan
  - Hillsborough, New Jersey
  - New York, New York
  - San Antonio, Texas
- Australia (2):
  - Fitzroy, South Australia
  - Melbourne, Victoria
- Canada (2):
  - Vancouver, British Columbia
  - Toronto, Ontario
- Montpellier, France
- New Zealand (2):
  - Auckland
  - Christchurch
- Poland (4):
  - Chorzów
  - Mysłowice
  - Warsaw
  - Wroclaw
- Bratislava, Slovakia